CLINICAL TRIAL: NCT03688217
Title: The Philani Mobile Video Intervention for Exclusive Breastfeeding (MOVIE) Study: a Cluster-randomized Controlled Trial of a Mobile Video Entertainment-education Intervention to Promote Exclusive Breastfeeding in South Africa
Brief Title: The Philani Mobile Video Intervention for Exclusive Breastfeeding (MOVIE) Study
Acronym: MOVIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles G. Prober (Other)
Collaborators: Heidelberg University (Other); University of Stellenbosch (Other); University of Cape Town (Other); Stanford University (Other)
Responsible Party: Sponsor-Investigator, Charles G. Prober, Founding Executive Director, Stanford Center for Health Education, Senior Associate Vice Provost for Health Education, Co-Senior Author, Professor of Pediatrics Microbiology and Immunology, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 46667
Record Dates: First submitted 2018-09-13; First posted 2018-09-28 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Exclusive Breastfeeding; Infant Feeding Practices
Keywords: exclusive breastfeeding; health education; entertainment-education; low- and middle-income countries; video-based; narrative; community-based
MeSH Terms: conditions — Breast Feeding; Health Education; Narration

STUDY DESIGN:
Intervention Model Description: This is a cluster-randomized controlled trial with baseline covariate adjustment and stratification.The randomization unit is the mentor-mother. The clusters are pregnant participants enrolled by each mentor-mother over the course of the trial. The randomization will be stratified by neighborhood type, to ensure balance of intervention versus control assignment by this covariate. The following baseline characteristics will be measured and adjusted for in the main analysis of the primary and secondary outcomes to increase statistical efficiency: 1. participant's number of previous children, 2. participant's age, 3. running water in the home, 4. electricity in the home, 5. participant's employment status, 6. participant's education level
Who Masked: Outcomes Assessor
Masking Description: Since data will be entered directly into a tablet device by the participant, the outcomes assessor (ie: the tablet) will have no knowledge of the interventions assigned to individual participants. Additionally, the phone survey company performing the follow-up surveys will be blinded to the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Philani Intervention Model+MOVIE (PIM+M) (Experimental): Participants will receive the standard PIM perinatal home visiting program together with the MOVIE intervention (13 entertainment-education videos about infant feeding). The PIM is a structured program of antenatal and postnatal home-visits covering foundational health promotion topics including nutrition in pregnancy, infant feeding, newborn care and maternal mental health among others. The MOVIE videos will be integrated into the regular home visiting program.
  Interventions: Behavioral: Philani Intervention Model+MOVIE (PIM+M)
- Philani Intervention Model (PIM) (Active Comparator): Participants will receive the standard PIM perinatal home visiting program, which is a structured program of antenatal and postnatal home-visits covering foundational health promotion topics including nutrition in pregnancy, infant feeding, newborn care and maternal mental health among others.
  Interventions: Behavioral: Philani Intervention Model (PIM)

INTERVENTIONS:
Behavioral: Philani Intervention Model+MOVIE (PIM+M) — The PIM+M intervention will involve the integration of the mobile video intervention into the standard perinatal counseling program offered by the intervention mentor-mothers. MOVIE intervention videos are narrated in English and isiXhosa, the languages spoken most widely among the study participants. Teaching videos are short (2-5 min.) and use simple language, avoiding medical jargon. The modularity of the videos facilitates delivery in any order and thus, they can be deployed at the discretion of each skilled mentor-mother, such that the health messages delivered are aligned with the individual needs of each participant at each perinatal stage. All videos will be administered at least once to each participant in the intervention group during the study period.
  Arms: Philani Intervention Model+MOVIE (PIM+M)
Behavioral: Philani Intervention Model (PIM) — The Philani Intervention Model (PIM) describes a structured program of antenatal and postnatal home-visits covering foundational health promotion topics including nutrition in pregnancy, infant feeding, newborn care and maternal mental health among others.
  Arms: Philani Intervention Model (PIM)

SUMMARY:
This cluster-randomized controlled trial seeks to evaluate the impact of a mobile video intervention for exclusive breastfeeding (MOVIE) on the infant feeding practices of mothers living in under-resourced communities in the Western Cape, South Africa. The trial will compare infant feeding practices in two groups of participants, enrolled in the Philani Mentor-Mother Outreach Program, a home-visiting program focused on community-based health promotion through peer-to-peer counseling. The participants in the intervention arm will receive the Philani Intervention Model (PIM), a perinatal health promotion intervention, together with the additional mobile, video intervention for exclusive breastfeeding. The participants in the control arm will receive only the standard PIM. Participants will be exposed to either the intervention or the control condition during pregnancy and the first five months after delivery. The central hypothesis in this trial is that, when compared with the control group, infant feeding practices in the intervention group will be significantly better aligned with current World Health Organization recommendations, after exposure to the Philani MOVIE intervention. The primary outcomes in this study are short-term exclusive breastfeeding, in the first month of life, and long-term exclusive breastfeeding, in the fifth month of life, (based on maternal 24-hour recall). Secondary outcomes include other infant feeding practices, such as early initiation of breastfeeding, any breastfeeding in the first month and in the fifth month of life, bottle-feeding, early introduction of complementary foods in the first month and in the fifth month of life and maternal knowledge in the first month and the fifth month post delivery.

DETAILED DESCRIPTION:
Background

The health benefits of exclusive breastfeeding (EBF), especially in low- and middle-income countries (LMIC), have been well documented. These include protection against infectious diseases, improved measures of intelligence and decreased risk of becoming overweight and developing diabetes. Globally, EBF could save the lives of an estimated 823 000 children under the age of five each year. Yet, despite World Health Organization recommendations that children should be exclusively breastfed for the first six months of life, EBF rates hover at only 37% in LMIC.

South Africa has one of the lowest rates of EBF in the world. Estimates of EBF rates under six months in South Africa range from 8% to the most generous estimate, 32% reported in the South Africa Demographic and Health Survey 2016. The health problems that result are largely due to unsafe formula feeding and the widespread practice of introducing solid foods early (often before three months) into the infant's diet. In South Africa, more than 70% of infants are given solid foods before reaching six months, the recommended age for initiating complementary feeding. Unsafe formula feeding and early introduction of solid foods can lead to diarrheal disease from pathogens entering the gut, as well as nutrient deficiencies when the foods introduced displace breastmilk without providing adequate nutrient density. The limited availability of reliable national data on infant feeding in South Africa complicates the design and evaluation of infant feeding interventions. However, systematic reviews of the literature suggest that large-scale interventions focused on educating mothers can increase the prevalence of EBF and decrease infant mortality.

Narrative, entertainment-education (E-E) approaches to health education have emerged as potentially powerful strategies for promoting positive health behavior change. E-E involves the delivery of health messages by embedding them in an entertainment media framework. A substantial body of research suggests that E-E is an effective way of influencing beliefs, attitudes and behaviors. The characteristics of particularly impactful E-E media include: a) appealing narratives, b) high-quality production, c) persuasive messages that are unobtrusive and d) high potential for involvement or identification with the presenters or characters portrayed. While E-E can take many forms, a video-based approach readily supports the optimized integration of these characteristics.

Video-based content, optimized for mobile devices, may also facilitate broad dissemination of health education, especially as the global penetration of mobile technology increases. Recent advances in mobile health (mHealth) messaging have already begun to facilitate the delivery of health messages at scale and researchers are increasingly recognizing the potential for mobile phones and tablets to play an important role in health education interventions in LMIC. South Africa is an example of a LMIC at the forefront of mHealth initiatives, due to its rapidly expanding penetration of mobile phones. National, maternal-child mHealth initiatives built around free, text-based messaging have attracted global attention and been well received. General "tech-savviness" in South Africa continues to grow, with 37% of adults reporting "smartphone" ownership and 42% reporting daily internet usage in 2016. Active experimentation with "WhatsApp", a widely used mobile communication tool that supports the transfer of videos, is also underway in many sectors, including health.

Even for South Africans who do not yet have access to mobile phones, a feasible dissemination pathway lies in the delivery of educational videos by community health workers (CHWs) who bring teaching tablets to their in-home counseling sessions. Numerous interventions that support women in their homes have demonstrated efficacy in improving breastfeeding rates. The Philani Maternal Child Health and Nutrition Trust is an example of a successful community based organization, employing "mentor-mothers", CHWs who offer in-home health promotion counseling to pregnant women and mothers within their communities. Data from both case studies and quantitative research suggest additional improvements in breastfeeding rates when synergistic interventions - for example, mass media interventions - are used to supplement successful community-based ones. Developing interventions that boost the efficacy of successful community-based programs represents a critical step towards ending preventable child and maternal deaths by 2030 (as called for by the World Health Organization (WHO) and UNICEF. Prior research in South Africa suggests that such synergistic interventions are even more effective when they are created in close collaboration with community-based programs, actively involving local stakeholders in the content creation process.

Aims

This study will achieve the following specific research aims: To establish the

1. Effectiveness of the Philani MOVIE intervention for improving exclusive breastfeeding practices among study participants
2. Effectiveness of the Philani MOVIE intervention for improving other infant feeding practices, and maternal knowledge among the study participants

Methods

A cluster-randomized controlled trial will be used to measure the effects of the Philani MOVIE intervention on infant feeding behaviors. Eighty-four mentor mothers will be randomized 1:1 into intervention and control arms, stratified by neighborhood type. Mentor-mothers in the control arm will provide the usual Philani Intervention Model (PIM) perinatal in-home counseling. Mentor-mothers in the intervention arm will provide standard care plus the MOVIE intervention (PIM+M). Based on sample size calculations described below, at least 1008 pregnant women will be enrolled in the study and mother-child pairs will be followed until five months of age. Cluster randomization will be done by a third party who is not employed by Philani, nor an in-country member of the research team.

Intervention

The Philani MOVIE intervention consists of 13 short, (2-5 min.), videos conveying current WHO infant feeding recommendations, the health rationale for these recommendations, historical information on global breastfeeding trends and contemporary challenges facing breastfeeding mothers. The intervention uses a narrative, entertainment-education approach, incorporating the personal stories of six South African mothers, three celebrities and three community mothers, alongside animations, illustrations and voiceovers by local South African voice talent.

Sample size calculation

The sample size calculation in this trial was based on the primary outcomes: exclusive breastfeeding in the first month and in the fifth month of life. Calculations were performed using standard methods for cluster-randomized controlled trials with baseline covariate adjustment and stratification. The randomization units were the mentor-mothers. An intra-cluster correlation of 0.1 was assumed for the two primary outcomes. Routine program data describing the performance of the 84 mentor-mothers participating in this trial was used to inform the power calculation. Based on this data, and a range of other data sources on breastfeeding in South Africa the investigators assumed that 40% of mothers exclusively breastfed their infants in the first month of life and 10% of mothers exclusively breastfed their infants in the fifth month of life. Assuming a correlation between the baseline measurements and the primary outcome of 0.30 and an average enrollment of 12 pregnant women per mentor-mother over the course of this study, the investigators estimated that the trial would have 80% power to detect at a 5% significance level a 13-percentage point increase in the primary outcome in the first month of life and a 9-percentage point increase in the primary outcome in the fifth month of life. This minimal detectable difference met the investigators' condition for policy relevance (an improvement of more than 15 percentage points). The total sample size was thus set for outcome assessment at 840 pregnant women plus 20% (to allow for loss to follow-up), i.e. 1008 pregnant women.

Data collection and training

Data will be collected via two tablet-based questionnaires, one in the first month post-delivery and the second in the fifth month post-delivery. Both questionnaires will be completed directly on the tablets by the participants and will include visual and audio prompts to overcome literacy barriers. Each of these surveys will be followed within one week by a telephone survey, administered by a professional phone survey research company, and will be used to verify the responses recorded on the tablet-based surveys and gather additional data on specific complementary foods introduced and on maternal knowledge.

Mentor-mothers in both the intervention and control groups will undergo training on basic research procedures. In total, six groups of ~15 mentor-mothers will attend a one-day training workshop over a one-week period, followed by a half-day refresher training workshop within three weeks of the first training. The workshops will include training on informed consent procedures, ethical principles, and the use of tablet devices to collect data on infant feeding practices. Mentor-mothers will be trained to open the questionnaires on the tablet and administer a practice questionnaire with the participant to ensure that the participant is comfortable and competent in working with the tablet. Once the mentor-mother is confident in the participant's ability to work with the tablet, they will hand it to the participants to complete the questionnaires independently, without input from their mentor-mother.

Mentor-mothers in both intervention and control groups will be afforded the opportunity to troubleshoot any concerns related to the use of the tablets or the research procedures for the duration of the study.

Mentor-mothers in the intervention group will undergo separate training sessions aimed at familiarizing them with the content of the Philani MOVIE intervention as well as allowing them to practice integrating the intervention into their existing perinatal home-visiting program. These training sessions will include role play activities, followed by feedback from peers and training facilitators.

Data Analysis

The primary analysis will be based on intention-to-treat at the unit of the individual newborn/individual mother, with standard errors adjusted for clustering at the level of the unit of randomization, i.e. the mentor-mothers. The investigators will adjust for baseline neighborhood type in addition to six additional baseline covariates detailed in the study design description. Mixed-effects generalized linear models will be used for the primary analysis, using a fixed effect for the assignment to treatment vs. control arm and a random effect for mentor-mother. In particular, the investigators will use modified Poisson models (generalized linear models with Poisson distribution and a logarithmic link function), for the binary outcomes, i.e., the primary outcomes as well as secondary outcomes, 3-13. Modified Poisson models were chosen because they generate estimates of risk ratios (and thus avoid the well-known interpretational difficulties associated with odds ratios) and because they converge more easily than alternative models that generate risk ratios (such as binomial models). For the continuous secondary outcomes (14 and 15), generalized linear models will be used with Gaussian distribution and identity link function.

ELIGIBILITY:
Inclusion Criteria:

* consenting pregnant clients, 20-40 weeks pregnant
* at least 18 years of age
* living within the catchment areas of the 84 mentor-mother CHWs taking part in this study
* enrolled in the Philani Mentor Mother Outreach Program

Exclusion Criteria:

* non-pregnant
* younger than 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1504 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Short-term Exclusive Breastfeeding (24-hour recall) | Measured at 1 month post-delivery via tablet based survey AND independent verification phone survey within one week
  Infant, age 1 month, was exclusively breastfed in the past 24 hours, per maternal report
Long-term Exclusive Breastfeeding (24-hour recall) | Measured at 5 months post-delivery via tablet based survey AND independent verification phone survey within one week
  Infant, age 5 months, was exclusively breastfed in the past 24 hours, per maternal report

SECONDARY OUTCOMES:
Short-term Exclusive Breastfeeding (since birth recall) | Measured at 1 month post-delivery via tablet based survey AND independent verification phone survey within one week
  Infant, age 1 month, was exclusively breastfed since birth, per maternal report
Long-term Exclusive Breastfeeding (since birth recall) | Measured at 5 months post-delivery via tablet based survey AND independent verification phone survey within one week
  Infant, age 5 months, was exclusively breastfed since birth, per maternal report
Early initiation of breastfeeding | Measured at 1 month post-delivery via tablet based survey AND independent verification phone survey within one week
  Infant was breastfed within the first hour of life (based on maternal recall)
Any breastfeeding at 1 month | Measured at 1 month post-delivery via tablet based survey AND independent verification phone survey within one week
  Infant, age 1 month, received any breastmilk in the past 24 hours, even if not exclusively breastfed
Any breastfeeding at 5 months | Measured at 5 months post-delivery via tablet based survey AND independent verification phone survey within one week
  Infant, age 5 months, received any breastmilk in the past 24 hours, even if not exclusively breastfed
Bottle-feeding at 1 month | Measured at 1 month post-delivery via tablet based survey AND independent verification phone survey within one week
  Infant, age 1 month, was fed using a bottle with a nipple in the past 24 hours
Bottle-feeding at 5 months | Measured at 5 months post-delivery via tablet based survey AND independent verification phone survey within one week
  Infant, age 5 months, was fed using a bottle with a nipple in the past 24 hours
Early introduction of complementary foods at 1 month (24-hour recall) | Measured at 1 month post-delivery by phone survey
  Infant, age 1 month, received complementary foods in the past 24 hours
Early introduction of complementary foods at 5 months (24-hour recall) | Measured at 5 months post-delivery by phone survey
  Infant, age 5 months, received complementary foods in the past 24 hours
Early introduction of complementary foods at 1 month (since birth recall) | Measured at 1 month post-delivery by phone survey
  Infant, age 1 month, received complementary foods at some point since birth
Early introduction of complementary foods at 5 months (since birth recall) | Measured at 5 months post-delivery by phone survey
  Infant, age 5 months, received complementary foods at some point since birth
Maternal knowledge at 1 month post-delivery | Measured at 1 month post-delivery by phone survey
  Short-term maternal knowledge of breastfeeding current recommendations and basic health principles relevant to infant feeding
Maternal knowledge at 5 months post-delivery | Measured at 5 months post-delivery by phone survey
  Long-term maternal knowledge of breastfeeding current recommendations and basic health principles

CONTACTS AND LOCATIONS:
Overall Officials: Maya Adam, MD, Principal Investigator — Stanford University; Till Bärnighausen, MD, ScD, Principal Investigator — Heidelberg University; Charles Prober, MD, Principal Investigator — Stanford University; Mark Tomlinson, PhD, Principal Investigator — University of Stellenbosch; Amnesty E LeFevre, PhD, Principal Investigator — University of Cape Town; Shannon McMahon, PhD, Principal Investigator — Heidelberg University
Locations (1):
- Philani Maternal Child Health and Nutrition Trust, Khayelitsha, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Background] Rollins NC, Bhandari N, Hajeebhoy N, Horton S, Lutter CK, Martines JC, Piwoz EG, Richter LM, Victora CG; Lancet Breastfeeding Series Group. Why invest, and what it will take to improve breastfeeding practices? Lancet. 2016 Jan 30;387(10017):491-504. doi: 10.1016/S0140-6736(15)01044-2. PMID 26869576
- [Background] Doherty T, Sanders D, Jackson D, Swanevelder S, Lombard C, Zembe W, Chopra M, Goga A, Colvin M, Fadnes LT, Engebretsen IM, Ekstrom EC, Tylleskar T; PROMISE EBF study group. Early cessation of breastfeeding amongst women in South Africa: an area needing urgent attention to improve child health. BMC Pediatr. 2012 Jul 24;12:105. doi: 10.1186/1471-2431-12-105. PMID 22827969
- [Background] Du Plessis L, Peer N, English R, Honikman S. Breastfeeding in South Africa: are we making progress? South African Health Review. 2016;2016(1):109-23.
- [Background] Cohen RJ, Brown KH, Canahuati J, Rivera LL, Dewey KG. Effects of age of introduction of complementary foods on infant breast milk intake, total energy intake, and growth: a randomised intervention study in Honduras. Lancet. 1994 Jul 30;344(8918):288-93. doi: 10.1016/s0140-6736(94)91337-4. PMID 7914260
- [Background] Kimmons JE, Dewey KG, Haque E, Chakraborty J, Osendarp SJ, Brown KH. Low nutrient intakes among infants in rural Bangladesh are attributable to low intake and micronutrient density of complementary foods. J Nutr. 2005 Mar;135(3):444-51. doi: 10.1093/jn/135.3.444. PMID 15735076
- [Background] Haroon S, Das JK, Salam RA, Imdad A, Bhutta ZA. Breastfeeding promotion interventions and breastfeeding practices: a systematic review. BMC Public Health. 2013;13 Suppl 3(Suppl 3):S20. doi: 10.1186/1471-2458-13-S3-S20. Epub 2013 Sep 17. PMID 24564836
- [Background] Chapman DJ, Morel K, Anderson AK, Damio G, Perez-Escamilla R. Breastfeeding peer counseling: from efficacy through scale-up. J Hum Lact. 2010 Aug;26(3):314-26. doi: 10.1177/0890334410369481. PMID 20715336
- [Background] Imdad A, Yakoob MY, Bhutta ZA. Effect of breastfeeding promotion interventions on breastfeeding rates, with special focus on developing countries. BMC Public Health. 2011 Apr 13;11 Suppl 3(Suppl 3):S24. doi: 10.1186/1471-2458-11-S3-S24. PMID 21501442
- [Background] Lumbiganon P, Martis R, Laopaiboon M, Festin MR, Ho JJ, Hakimi M. Antenatal breastfeeding education for increasing breastfeeding duration. Cochrane Database Syst Rev. 2016 Dec 6;12(12):CD006425. doi: 10.1002/14651858.CD006425.pub4. PMID 27922724
- [Background] Hinyard LJ, Kreuter MW. Using narrative communication as a tool for health behavior change: a conceptual, theoretical, and empirical overview. Health Educ Behav. 2007 Oct;34(5):777-92. doi: 10.1177/1090198106291963. Epub 2006 Dec 15. PMID 17200094
- [Background] Slater MD, Rouner D. Entertainment-education and elaboration likelihood: Understanding the processing of narrative persuasion. Communication Theory. 2002;12(2):173-91.
- [Background] Rogers EM, Vaughan PW, Swalehe RM, Rao N, Svenkerud P, Sood S. Effects of an entertainment-education radio soap opera on family planning behavior in Tanzania. Stud Fam Plann. 1999 Sep;30(3):193-211. doi: 10.1111/j.1728-4465.1999.00193.x. PMID 10546311
- [Background] Shen F, Han J. Effectiveness of entertainment education in communicating health information: A systematic review. Asian Journal of Communication. 2014;24(6):605-16.
- [Background] Wilson KE, Beck VH. Entertainment outreach for women's health at CDC. J Womens Health Gend Based Med. 2002 Sep;11(7):575-8. doi: 10.1089/152460902760360522. No abstract available. PMID 12396890
- [Background] Aranda-Jan CB, Mohutsiwa-Dibe N, Loukanova S. Systematic review on what works, what does not work and why of implementation of mobile health (mHealth) projects in Africa. BMC Public Health. 2014 Feb 21;14:188. doi: 10.1186/1471-2458-14-188. PMID 24555733
- [Background] Gurman TA, Rubin SE, Roess AA. Effectiveness of mHealth behavior change communication interventions in developing countries: a systematic review of the literature. J Health Commun. 2012;17 Suppl 1:82-104. doi: 10.1080/10810730.2011.649160. PMID 22548603
- [Background] Sondaal SF, Browne JL, Amoakoh-Coleman M, Borgstein A, Miltenburg AS, Verwijs M, Klipstein-Grobusch K. Assessing the Effect of mHealth Interventions in Improving Maternal and Neonatal Care in Low- and Middle-Income Countries: A Systematic Review. PLoS One. 2016 May 4;11(5):e0154664. doi: 10.1371/journal.pone.0154664. eCollection 2016. PMID 27144393
- [Background] World Health Organization. mHealth: New horizons for health through mobile technologies: second global survey on eHealth. 2011. Geneva: WHO Google Scholar. 2014.
- [Background] Labrique AB, Vasudevan L, Kochi E, Fabricant R, Mehl G. mHealth innovations as health system strengthening tools: 12 common applications and a visual framework. Glob Health Sci Pract. 2013 Aug 6;1(2):160-71. doi: 10.9745/GHSP-D-13-00031. eCollection 2013 Aug. PMID 25276529
- [Background] Kallander K, Tibenderana JK, Akpogheneta OJ, Strachan DL, Hill Z, ten Asbroek AH, Conteh L, Kirkwood BR, Meek SR. Mobile health (mHealth) approaches and lessons for increased performance and retention of community health workers in low- and middle-income countries: a review. J Med Internet Res. 2013 Jan 25;15(1):e17. doi: 10.2196/jmir.2130. PMID 23353680
- [Background] Diamond L. Liberation technology. In Search of Democracy: Routledge; 2015. p. 148-62.
- [Background] Kakihara M, editor Grasping a Global View of Smartphone Diffusion: An Analysis from a Global Smartphone Study. ICMB; 2014.
- [Background] Kreutzer T. Generation mobile: online and digital media usage on mobile phones among low-income urban youth in South Africa. Retrieved on March. 2009;30(2009):903-20.
- [Background] Barron P, Pillay Y, Fernandes A, Sebidi J, Allen R. The MomConnect mHealth initiative in South Africa: Early impact on the supply side of MCH services. J Public Health Policy. 2016 Nov;37(Suppl 2):201-212. doi: 10.1057/s41271-016-0015-2. PMID 27899795
- [Background] Seebregts C, Barron P, Tanna G, Benjamin P, Fogwill T. MomConnect: an exemplar implementation of the health normative standards framework in South Africa. South African Health Review. 2016;2016(1):125-35.
- [Background] Poushter J. Smartphone ownership and internet usage continues to climb in emerging economies. Pew Research Center. 2016;22.
- [Background] Shambare R. The adoption of WhatsApp: Breaking the vicious cycle of technological poverty in South Africa. Journal of economics and behavioral studies. 2014;6(7):542.
- [Background] Anstey Watkins JOT, Goudge J, Gomez-Olive FX, Griffiths F. Mobile phone use among patients and health workers to enhance primary healthcare: A qualitative study in rural South Africa. Soc Sci Med. 2018 Feb;198:139-147. doi: 10.1016/j.socscimed.2018.01.011. Epub 2018 Jan 10. PMID 29335160
- [Background] Coetzee B, Kohrman H, Tomlinson M, Mbewu N, Le Roux I, Adam M. Community health workers' experiences of using video teaching tools during home visits-A pilot study. Health Soc Care Community. 2018 Mar;26(2):167-175. doi: 10.1111/hsc.12488. Epub 2017 Sep 5. PMID 28872210
- [Background] Tomlinson M, Rotheram-Borus MJ, le Roux IM, Youssef M, Nelson SH, Scheffler A, Weiss RE, O'Connor M, Worthman CM. Thirty-Six-Month Outcomes of a Generalist Paraprofessional Perinatal Home Visiting Intervention in South Africa on Maternal Health and Child Health and Development. Prev Sci. 2016 Nov;17(8):937-948. doi: 10.1007/s11121-016-0676-x. PMID 27438294
- [Background] Black RE, Taylor CE, Arole S, Bang A, Bhutta ZA, Chowdhury AMR, Kirkwood BR, Kureshy N, Lanata CF, Phillips JF, Taylor M, Victora CG, Zhu Z, Perry HB. Comprehensive review of the evidence regarding the effectiveness of community-based primary health care in improving maternal, neonatal and child health: 8. summary and recommendations of the Expert Panel. J Glob Health. 2017 Jun;7(1):010908. doi: 10.7189/jogh.07.010908. PMID 28685046
- [Background] Mosavel M, Simon C, van Stade D, Buchbinder M. Community-based participatory research (CBPR) in South Africa: engaging multiple constituents to shape the research question. Soc Sci Med. 2005 Dec;61(12):2577-87. doi: 10.1016/j.socscimed.2005.04.041. Epub 2005 Jun 13. PMID 15955605
- [Background] World Health Organization. Indicators for assessing infant and young child feeding practices. Part I: definition. Geneva: 2008.
- [Background] Use CfMPfH. Guideline on adjustment for baseline covariates. European Medicines Agency; 2014.
- [Background] Barnhart D, Hertzmark E, Liu E, Mungure E, Muya AN, Sando D, Chalamilla G, Ulenga N, Barnighausen T, Fawzi W, Spiegelman D. Intra-Cluster Correlation Estimates for HIV-related Outcomes from Care and Treatment Clinics in Dar es Salaam, Tanzania. Contemp Clin Trials Commun. 2016 Dec 15;4:161-169. doi: 10.1016/j.conctc.2016.09.001. Epub 2016 Sep 14. PMID 27766318
- [Background] Goga AE, Doherty T, Jackson DJ, Sanders D, Colvin M, Chopra M, Kuhn L. Infant feeding practices at routine PMTCT sites, South Africa: results of a prospective observational study amongst HIV exposed and unexposed infants - birth to 9 months. Int Breastfeed J. 2012 Apr 3;7:4. doi: 10.1186/1746-4358-7-4. PMID 22472507
- [Derived] Adam M, Johnston J, Job N, Dronavalli M, Le Roux I, Mbewu N, Mkunqwana N, Tomlinson M, McMahon SA, LeFevre AE, Vandormael A, Kuhnert KL, Suri P, Gates J, Mabaso B, Porwal A, Prober C, Barnighausen T. Evaluation of a community-based mobile video breastfeeding intervention in Khayelitsha, South Africa: The Philani MOVIE cluster-randomized controlled trial. PLoS Med. 2021 Sep 28;18(9):e1003744. doi: 10.1371/journal.pmed.1003744. eCollection 2021 Sep. PMID 34582438
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] Adam M, Tomlinson M, Le Roux I, LeFevre AE, McMahon SA, Johnston J, Kirton A, Mbewu N, Strydom SL, Prober C, Barnighausen T. The Philani MOVIE study: a cluster-randomized controlled trial of a mobile video entertainment-education intervention to promote exclusive breastfeeding in South Africa. BMC Health Serv Res. 2019 Apr 2;19(1):211. doi: 10.1186/s12913-019-4000-x. PMID 30940132